CLINICAL TRIAL: NCT04978662
Title: Determination of Sleep Disorder and Chronotype in Children and Adolescents With Type 1 Diabetes; Observation of the Impact on Glycemic Control and Treatment
Brief Title: Sleep and Chronotype in Children With Type 1 Diabetes
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Marmara University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Perran Boran, Professor of Pediatrics, Marmara University
Other Study IDs: 120S789
Record Dates: First submitted 2021-07-06; First posted 2021-07-27 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Mellitus, Type 1; sleep; adolescent; actigraphy; blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Type 1 diabetes is the most common metabolic disorder in children and adolescents. Sleep is important for prognosis and several sleep parameters are related to metabolic control. However, limited number of studies in children and adolescents showed mixed results and recommendations about how to address sleep in the clinical care of diabetes in children are still lacking. There is a need to examine the potential role of sleep in developing preventive interventions for diabetes management in children and adolescents.

The authors aimed to describe sleep/wake patterns ,sleep problems, and chronotype of children and adolescents with type 1 diabetes, and to assess the relation of sleep measures with metabolic control and treatment.

The study has a prospective observational cross-sectional design. An estimated sample size is calculated as 83. Children diagnosed with type 1 diabetes between 6 to 18 years of age will be recruited from two pediatric endocrinology centers specialized in diabetes. Sleep/wake pattern will be assessed by actigraphy, and sleep diaries. Sleep disorder will be assessed by the Diagnostic and Statistical Manual for Mental Disorders (DSM-5) Sleep Disorder Scale, and Chronotype Questionnaire will be used to determine the chronotype.

DETAILED DESCRIPTION:
Type 1 diabetes is the most common metabolic disorder in children and adolescents. Sleep is important for prognosis and several sleep parameters are related to metabolic control. However, limited number of studies in children and adolescents showed mixed results and recommendations about how to address sleep in the clinical care of diabetes in children are still lacking. There is a need to examine the potential role of sleep in preventive interventions.

The authors aimed to describe sleep/wake patterns ,sleep problems, and chronotype of children and adolescents with type 1 diabetes, and to assess the relation of sleep measures with metabolic control and treatment.

The study has a prospective observational cross-sectional design. An estimated sample size is calculated as 83. Children diagnosed with type 1 diabetes between 6 to 18 years of age will be recruited from two pediatric endocrinology centers specialized in diabetes. Sleep/wake pattern will be assessed by actigraphy, and sleep diaries. Sleep wake patterns will be assessed by Philips Respironics Mini-Mitter Actiwatch-2 for at least 3 days at home environment and sleep diaries within 5-minute intervals will be filled out by parents. Actigraphy is a validated wristwatch-like device that distinguishes sleep from wakefulness based on accelerometer measured movement.

Sleep disorder will be assessed by the Diagnostic and Statistical Manual for Mental Disorders (DSM-5) Sleep Disorder Scale, and Chronotype Questionnaire will be used to determine the chronotype.

For metabolic control, targeted standard values will be used for continuous glucose measurement. (Target daily blood glucose ranges 70-180 mg/dl, <4% <70 mg/dl, <1% <54 mg/dl, <25% >180 mg/dl, <5% rate >250 mg/dl). The latest Hemoglobin A1c level will also be evaluated.

A questionnaire developed by the investigators including sociodemographic characteristics, and diabetes related information will be gathered from the patient records.

ELIGIBILITY:
Inclusion Criteria:

* aged between 6 to 18 years
* use of continuous glucose monitoring system

Exclusion Criteria:

* acute medical condition that can impact sleep (diabetes keto acidosis, cold, influenza)
* diagnosed neurodevelopmental or behavioral condition like autism spectrum disorder or Attention Deficit/Hyperactivity Disorder
* diagnosed sleep disorder (Obstructive Sleep Apnea)
* Current use of medications that can impact sleep (diphenhydramine)

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents diagnosed with Type 1 Diabetes aged between 6 to 18 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-07-06 (Actual); Primary Completion 2021-10 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
sleep wake patterns measured by actigraphy | baseline
  sleep wake patterns
sleep disorder | Baseline
  sleep disorder measured with the Diagnostic and Statistical Manual for Mental Disorders (DSM-5) Sleep Disorder Scale. The scale has an 8-item parent form, that could be filled up by parents or legal guardians of children aged between 6-17 years, and a 9-item self report form to be filled up by adolescents aged between 11-17 years. For each item, the caregiver is asked to rate the severity of symptoms related to sleep disorders that occurred within the past 7 days, she/he had observed in his/her child. The scale has a 5-point Likert type rating (1=never, 2=very little/rarely, 3=sometimes, 4=most of the time, 5=almost all the time). Total scores range between 8-40 and higher scores indicate presence of much more severe sleep-related problems.
chronotype | baseline
  chronotype measured with Chronotype Questionnaire.Children's Chronotype Questionnaire (CCTQ) is a parent report, 27-item mixed format questionnaire measuring chronotype of children in multiple domains : the midsleep point on free days (MSF), a morningness/eveningness scale(M/E) score, and a five-point chronotype (CT) score.

SECONDARY OUTCOMES:
metabolic control | baseline
  metabolic control measured by number of hypo and hyperglycemic episodes over the past month
metabolic control | baseline
  metabolic control measured by the most recent hemoglobin A1c
treatment | baseline
  treatment measured by insulin dose per kilogram

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No